CLINICAL TRIAL: NCT06335732
Title: Prevalenc Of Lumbosacral Radiculopathy Among Physiotherapists Of Pediatric Rehabilitation
Brief Title: Prevalenc Of Lumbosacral Radiculopathy Among Physiotherapists Of Pediatric Rehabilitation OF PEDIATRIC REHABILITATION
Status: Completed | Type: Observational
Sponsor: Kerolous Ishak Shehata (Other)
Responsible Party: Sponsor-Investigator, Kerolous Ishak Shehata, Prevalenc Of Lumbosacral Radiculopathy Among Physiotherapists Of Pediatric Rehabilitation, October 6 University
Organization: October 6 University (Other)
Other Study IDs: P.T.REC/012/004394
Record Dates: First submitted 2024-03-22; First posted 2024-03-28 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Prevalence, Lumbosacral Radiculopathy
Keywords: Prevalence, Lumbosacral radiculopathy, Low back pain.
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Cross section study; single group related measurement design. — Two hundred pediatric physiotherapists from both genders were participated in the current study. They were selected randomly from the Outpatient Clinic of pediatric physiotherapists of Hospitals of Ministry of Health in Cairo-Egypt, the duration of this study was six months started from December 2022 to June 2023

SUMMARY:
Determine the prevalence of lumbosacral radiculopathy among pediatric physiotherapists in the ministry of health in Cairo, Egypt.

DETAILED DESCRIPTION:
the aim of current study was to determine the prevalence of lumbosacral radiculopathy among pediatric physiotherapists in the ministry of health in Cairo, Egypt.

ELIGIBILITY:
Inclusion Criteria:

* a) The age of the subjects ranged from 25-40 years old; b) all subjects working in Ministry of Health in Cairo-Egypt; c) BMI <30

Exclusion Criteria:

* they were with history of bone disease, renal, liver or endocrinal disorders; b) having lumbosacral radiculopathy before working as pediatric physiotherapists, c) having trauma in back or accident and pregnant pediatric physiotherapists

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Two hundred pediatric physiotherapists from both genders were participated in the current study. They were selected randomly from the Outpatient Clinic of pediatric physiotherapists of Hospitals of Ministry of Health in Cairo-Egypt, the duration of this study was six months started from December 2022 to June 2023.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2022-12-05 (Actual); Primary Completion 2023-06-08 (Actual); Study Completion 2023-08-22 (Actual)

PRIMARY OUTCOMES:
The Roland-Morris disability scale (RMS) | up to 6 months
  The Roland-Morris disability scale (RMS) for disability secondary to low back pain is a validated and popular instrument in clinical22 practice,
Straight Leg Raising (SLR) | up to 6 months
  Straight Leg Raising (SLR) is widely used to diagnose lumbosacral nerve root irritation

CONTACTS AND LOCATIONS:
Locations (1):
- Kerolous Ishak Shehata, Cairo, Egypt